CLINICAL TRIAL: NCT02779517
Title: Mobile Service Robot for Task-Oriented Stroke Therapy: User Evaluations
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 819669
Record Dates: First submitted 2016-03-31; First posted 2016-05-20 (Estimated); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Stroke
Keywords: upper extremity; stroke; rehabilitation; robotics; telepresence; elderly; aged; Housing for the elderly; retirement; homes for the aged
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Focus groups- Patients: Subjects with or without an upper extremity disability will be asked to observe and interact with the mobile service robot.
  Interventions: Other: Mobile Service Robot Survey for Patients
- Focus Groups-clinicians: Clinicians with neuro-rehab experience.
  Interventions: Other: Mobile Service Robot Survey

INTERVENTIONS:
Other: Mobile Service Robot Survey — The goal is to build a low-cost mobile service robot that will focus on the simple, but key, repetitive, data-driven tasks that robots do well. Rather than attempt to create a robot helper that mimics humans, the goal is to free human caregivers from the time-consuming tasks that robots can accomplish with facility, thereby allowing humans to focus on tasks that humans do best (i.e. human contact).
  Groups: Focus Groups-clinicians
Other: Mobile Service Robot Survey for Patients — The goal is to build a low-cost mobile service robot that will focus on the simple, but key, repetitive, data-driven tasks that robots do well. Rather than attempt to create a robot helper that mimics humans, the goal is to free human caregivers from the time-consuming tasks that robots can accomplish with facility, thereby allowing humans to focus on tasks that humans do best (i.e. human contact). This survey differs in terms of design questions.
  Groups: Focus groups- Patients

SUMMARY:
By developing an affordable mobile service robot for therapeutic activities in a health center environment, this project addresses the issue of both the high cost and man-power required to provide rehabilitation for stroke survivors and other patients. Our goal is to measure users - clinician and patient - responses to a telepresence robot, VGo, that has been modified with a humanoid torso robot, NAO, to facilitate remote communication between the patient and clinician, and to complete supervisory exercise coaching.

DETAILED DESCRIPTION:
This is a short demonstration and survey study. Clinical staff and patients will be gathered together and our idea for the mobile service robot will discussed. A demonstration of the telepresence feature of the robots and the NAO robot greeting and helping them with simple exercises will follow (e.g., pick up and object that is handy and lift their hands over their heads). The approximately 30-minute demonstration part of the study will start with an introduction and explanation about the project and a short speech about the Rehabilitation and Robotics Lab. After the demonstration the oral consent will be read and surveys will be handed out to those study participants who agree to complete them; if necessary, the research team will assist the study participant with the survey. Surveys will then be collected, and the group will be thanked by the research team.

ELIGIBILITY:
Inclusion Criteria:

* Certified rehabilitation healthcare professionals
* Participants with upper extremity disabilities
* Participant must be older than 18 years

Exclusion Criteria:

-Less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Therapists with neuro-rehab experience. Patients with neural injury.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2014-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Perception of the interaction with the robot | up to 1 week
  Perception of the robot measured by surveys administered to participants as well as by observation with the robot.
Usability of the robot | up to 1 week
  Portability, ease of set up, cost, and appearance measured by surveys administered to participants as well as by observation with the robot.
Sociability with the robot | up to 1 week
  Sociability of robot measured by surveys administered to participants as well as by observation with the robot.

SECONDARY OUTCOMES:
Design requirements | up to 1 week
  Design requirements measured by surveys administered to participants as well as by observation with the robot.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle J Johnson, PhD, Principal Investigator — Penn Medicine Rittenhouse
Locations (1):
- Penn Medicine Rittenhouse, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilk R. and Johnson MJ. 5th IEEE RAS/EMBS International Conference on Biomedical Robotics and Biomechatronics. ; 08/2014. doi:10.1109/BIOROB.2014.6913816